CLINICAL TRIAL: NCT02409849
Title: Randomized Phase II Study of Octreotide LAR as Maintenance Treatment After First-line Chemotherapy for Patients With Unresectable or Metastatic Gastro-entero-pancreatic or Esophageal Neuroendocrine Carcinomas
Brief Title: Octreotide LAR as Maintenance Treatment for Patients With NEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, GI Oncology Department, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJT-NEC-002
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Gastro-entero-pancreatic Carcinoma; Esophageal Neuroendocrine Carcinoma
Keywords: Octreotide LAR; Neuroendocrine carcinomas; unresectable or metastatic; Disease-free survival
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention)
- Octreotide LAR treatment (Experimental): The patients with unresectable or metastatic GEP or esophageal NEC who got CR/PR/SD after chemotherapy with IP or EP regimen qualified with the inclusion criteria are enrolled. All the patients enrolled in our study will be randomly assigned to receive octreotide LAR (group A) as maintenance treatment or follow up (group B) to disease progression.
  Interventions: Drug: Octreotide lar

INTERVENTIONS:
Drug: Octreotide lar
  Other Names: Octreotide lar 30mg，deep i.m，q28d，
  Arms: Octreotide LAR treatment

SUMMARY:
This is phase II study on the efficacy of octreotide lar as maintenance treatment after first-line chemotherapy for patients with unresectable or metastatic gastro-entero-pancreatic or esophageal neuroendocrine carcinomas.

DETAILED DESCRIPTION:
This is a prospective, randomized, open label study on the efficacy of octreotide lar as maintenance treatment after first-line chemotherapy for patients with unresectable or metastatic gastro-entero-pancreatic or esophageal neuroendocrine carcinomas.The patients with unresectable or metastatic GEP or esophageal NEC who got CR/PR/SD after chemotherapy with IP or EP regimen qualified with the inclusion criteria are enrolled. All the patients enrolled in our study will be randomly assigned to receive octreotide LAR (group A) as maintenance treatment or follow up (group B) to disease progression. Treatment will be discontinued on withdrawal of patient consent, disease progression, unacceptable toxicity, a treatment delay of >2 weeks, or major protocol violations, after which patients were followed up every 3 months for a minimum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of high grade (poorly differentiated) gastro-entero-pancreatic neuroendocrine carcinoma.
2. High grade neuroendocrine carcinoma of esophageal or unknown primary site (if a pulmonary primary has been excluded)
3. Metastatic or unresectable disease
4. Measurable disease
5. Accepted chemotherapy with EP or IP regimen for no less than three months
6. Effectiveness with CR/PR/SD
7. Informed consent
8. Performance status of 0 or 1
9. Adequate bone marrow function (defined as absolute neutrophil count [ANC] >= 1500, platelet count [PLT] >= 75,000 and a hemoglobin [Hgb] >= 9).
10. Adequate hepatic function with a bilirubin of <= 2.0 mg/dl, and aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) <= 2.5 times the upper limits of normal, unless caused by liver metastasis. If caused by metastasis, then should be SGPT and SGOT <= 5 times the upper limits of normal.

Adequate renal function defined as serum creatinine <= 1.5 mg/dl.

Exclusion Criteria:

1. Patients who are on EP or IP chemotherapy for less than three months .
2. Effectiveness with PD.
3. Patients with brain metastases are not eligible.
4. Patients with New York Heart Association (NYHA) Class III or IV heart disease are not eligible as well as those patients with history of angina, myocardial infarction, or congestive heart failure within six months.
5. Pregnant or lactating women. All women of child bearing potential must have a negative pregnancy test prior to entry into the study. All patients of child bearing potential must be advised of the importance of avoiding pregnancy and using appropriate methods of contraception while participating in this investigational trial.
6. Patients with serious complicated infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
7. Patients with psychiatric disorders rendering them incapable of complying with the requirements of the protocol.
8. Patients with serum calcium > 12 mg/dl or symptomatic hypercalcemia under treatment.
9. Patients with osseous metastasis as only site of disease.
10. Patients with any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial.
11. Patients with known Gilbert's syndrome are ineligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-11 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years

SECONDARY OUTCOMES:
OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China